CLINICAL TRIAL: NCT03795090
Title: A Multi-level Antimicrobial Surface Coating for a Healthier Environment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hong Kong University of Science and Technology (Other)
Collaborators: Kowloon Hospital, Hong Kong (Other); Queen Elizabeth Hospital, Hong Kong (Other); Innovation and Technology Commission, Hong Kong (Other)
Responsible Party: Principal Investigator, King Lun Yeung, Professor, Hong Kong University of Science and Technology
Allocation: Non-Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ITT/008/15GP
Record Dates: First submitted 2018-11-28; First posted 2019-01-07 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Hospital Acquired Infections
Keywords: Antimicrobial coating, MDRO, MRSA, Patient Privacy Curtains

STUDY DESIGN:
Intervention Model Description: Phase 1, even numbers in coding are treatment and odd coded curtains are control (Blind) Phase 2, odd numbers in coding are treatment and even coded curtains are control (Blind) Phase 3, even numbers in coding are treatment and odd coded curtains are control (Blind)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study is complete blind as only principal investigator knows the coding on curtains and he can differentiate between two physically similar looking patient privacy curtains.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular Patient privacy curtain (Active Comparator): Control arm is a regular patient privacy curtain, washed and dried in hospital laundry using commercially available sodium hypochlorite and hydrogen peroxide.
  Interventions: Combination Product: Regular Patient privacy curtain
- Antimicrobial Coated Curtains (Experimental): Treatment arm is an antimicrobial coated curtains, which is obtained by dipping the hospital laundered curtains into the antimicrobial coating. The curtains are then dried and provided to the nursing/supporting staff.
  Interventions: Combination Product: Regular Patient privacy curtain; Combination Product: Antimicrobial Coated curtains

INTERVENTIONS:
Combination Product: Regular Patient privacy curtain — Laundered curtains, used in the hospital, coming from the hospital inventory.
Combination Product: Antimicrobial Coated curtains — Antimicrobial coating consist of active polymers that are approved by USFDA and USEPA.
  Arms: Antimicrobial Coated Curtains

SUMMARY:
This project aimed to study the use of the multi-level antimicrobial coating in a working hospital environment. Patient privacy curtains from a public sector hospital were coated and installed in rehabilitation ward in comparison of normally washed curtains in the same setting and compared the mean reduction on both control and treatment end to assess the effectiveness of coating against hospital acquired infections including multidrug resistant organisms (MDROs).

DETAILED DESCRIPTION:
1. A multi-level antimicrobial coating was produced in the Hong Kong University of Science and Technology (HKUST) laboratory using the newly developed staged flow micromixing to prepare contact-killing and anti-adhesion coating made of US-FDA approved polymeric materials. The process was optimized to scale-up the production to 5 liters per hour. 300 liters of the multi-level antimicrobial coating was prepared for the study for a total of 24 weeks as three liters of the coating was needed for one patient privacy curtain.
2. The study was conducted in the rehabilitation ward of the Kowloon Hospital including both male and female cubicles. It was carried out in three stages with each stage consisting of survey and a four weeks' observation period, separated by three weeks' washout period. In the rehabilitation ward of Kowloon Hospital, a set of male and female cubicle was recruited for the study after getting maximum number of bacterial contamination on patient privacy curtains in pilot study of 8 weeks. Each cubicle had 12 curtains besides admitted patients where all the samples are collected.
3. Environmental sampling was carried out using sponge swab on the surfaces of the patient privacy curtains. The total bacteria count and quantitative isolation of MRSA was done using established protocols. The total bacteria count provides a quantitative measure of surface cleanliness, while the methicillin-resistant Staphylococcus aureus (MRSA) count was indicative of the risk of contact transmission from contaminated surfaces. 2-4 weeks survey provided control data on the cleanliness of patients privacy curtains in terms of total bacteria and MRSA counts.

   During the study period, the Kowloon Hospital/Queen Elizabeth Hospital infection control team monitored MDROs regularly as part of their routine operation. The procedure and schedule was followed strictly the infection control protocol. All infection control measures implemented after isolation of MDROs were followed according to the hospital's usual practice as advised by the infection control team. In the study, the identification of the organisms in patients more than 48 hours after admission without prior isolation of the organisms in clinical or screening specimens was defined as nosocomial.
4. The investigators demonstrated a cross-over intervention study. In the first stage of study, half of the patient privacy curtains were considered as treatment (antimicrobial coated) and the other half of the curtains as control in the same setting in a cubicle. As the study was double blind, so coding was done to identify the treatment as control curtains.
5. Sample were taken from eight highly touched areas of 50x50 cm² on weekly bases for three consecutive weeks on 7th day of first installation. On each period/phase 480, 576 and 786 samples were collected accordingly using the developed sample protocol. In total, the investigators collected 1824 samples from 76 patient privacy curtains in which 912 (50%) were control curtain and 912 (50%) are antimicrobial coated curtains.
6. Healthcare workers from the participating wards were assessed for their acceptance of the multilevel antimicrobial disinfectant coating by way of a questionnaire. Additional reformulation may be necessary to increase the acceptability of the coating technology to the healthcare workers.
7. For the bacteria count, duplicate plates of tryptic soy agar (TSA) for total bacteria count and Chromagar MRSA (selective agar for MRSA detection) were used for enumeration. CFU/m² is calculated after 48 hours incubation at 37°C. Data was analyzed using Statistical Package for the Social Sciences (SPSS) V.25 to assess the effectiveness of the coating in reducing the contamination level of the surface. The total bacteria count on the patient privacy curtains was compared between the control and treatment group using Mann-Whitney test and T-test. ANOVA analysis allowed the comparison of different periods of study of phase wise as well as week wise. The significance of the statistical test is defined to have a P value <0.05.

ELIGIBILITY:
Inclusion Criteria:

* A convalescence ward with reasonable amount of nursing activities
* No recent history of outbreaks of communicable diseases in the wards

Exclusion Criteria:

* Wards with little nursing activities including infirmary wards
* Wards with frequent outbreaks which lead to excessive curtain changes

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change in total bacteria count and MRSA in control vs treatment patient privacy curtains | 12 weeks
  To quantify the effectiveness of antimicrobial coating, percentage change (both in log and linear scale) in mean bacterial count (CFU/m2 units) in control versus treatment curtains is used. The data was collected in 3 phases of 4 weeks each, so the time frame used is representative of the complete observation period.
Durability of antimicrobial coating in affecting bacterial load amongst treated patient privacy curtains | 12 weeks
  Change in bacterial load amongst treatment curtains is observed as a function of time during each phase of the data collection period (for 4 weeks). In total, data was collected in 3 phases of 4 weeks each, so the total observation period is 12 weeks and timeframe of each frame is 4 weeks.

SECONDARY OUTCOMES:
Agreement/disagreement of hospital staff regarding technology acceptance and adaptation | 4 weeks
  A survey was conducted using a self-structured questionnaire to get feedback from the hospital staff regarding their acceptance of the technology. The questionnaire contained questions regarding the physical (smell, appearance and feel) aspects of the coating as well as general approval/disapproval based on their experience with the technology. A scale of -5(worst) to +5(best), with 0 representing neutral was used, representing a dimensionless quantity based on staff's personal preferences. Mean of the user's response to each question was used for quantification. The users observed the technology during the entire 12 weeks of the study period (during all 3 phases of data collection). Users were give a 4-week time period to submit their survey responses.

CONTACTS AND LOCATIONS:
Overall Officials: King Lun Yeung, PhD, Principal Investigator — Hong Kong University of Science and Technology; Chritropher Lai, MBChB, FRCP, Study Chair — Kowloon Hospital; Dominic Tsang, MBChB, FRCP, Study Director — Kowloon Hospital
Locations (1):
- Kowloon Hospital, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
This is under discussion and final decision will be made later.

REFERENCES:
- [Background] Klein E, Smith DL, Laxminarayan R. Hospitalizations and deaths caused by methicillin-resistant Staphylococcus aureus, United States, 1999-2005. Emerg Infect Dis. 2007 Dec;13(12):1840-6. doi: 10.3201/eid1312.070629. PMID 18258033
- [Background] de Kraker ME, Davey PG, Grundmann H; BURDEN study group. Mortality and hospital stay associated with resistant Staphylococcus aureus and Escherichia coli bacteremia: estimating the burden of antibiotic resistance in Europe. PLoS Med. 2011 Oct;8(10):e1001104. doi: 10.1371/journal.pmed.1001104. Epub 2011 Oct 11. PMID 22022233
- [Background] Carling PC, Von Beheren S, Kim P, Woods C; Healthcare Environmental Hygiene Study Group. Intensive care unit environmental cleaning: an evaluation in sixteen hospitals using a novel assessment tool. J Hosp Infect. 2008 Jan;68(1):39-44. doi: 10.1016/j.jhin.2007.09.015. Epub 2007 Dec 11. PMID 18069083
- [Background] Huang SS, Datta R, Platt R. Risk of acquiring antibiotic-resistant bacteria from prior room occupants. Arch Intern Med. 2006 Oct 9;166(18):1945-51. doi: 10.1001/archinte.166.18.1945. PMID 17030826
- [Background] Datta R, Platt R, Yokoe DS, Huang SS. Environmental cleaning intervention and risk of acquiring multidrug-resistant organisms from prior room occupants. Arch Intern Med. 2011 Mar 28;171(6):491-4. doi: 10.1001/archinternmed.2011.64. PMID 21444840
- [Background] Otter JA, Yezli S, Perl TM, Barbut F, French GL. The role of 'no-touch' automated room disinfection systems in infection prevention and control. J Hosp Infect. 2013 Jan;83(1):1-13. doi: 10.1016/j.jhin.2012.10.002. Epub 2012 Nov 26. PMID 23195691
- [Background] Carling PC, Parry MM, Rupp ME, Po JL, Dick B, Von Beheren S; Healthcare Environmental Hygiene Study Group. Improving cleaning of the environment surrounding patients in 36 acute care hospitals. Infect Control Hosp Epidemiol. 2008 Nov;29(11):1035-41. doi: 10.1086/591940. PMID 18851687

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-02): https://cdn.clinicaltrials.gov/large-docs/90/NCT03795090/Prot_SAP_000.pdf